CLINICAL TRIAL: NCT01611948
Title: Pharmacological Treatment of Cannabis Withdrawal and Dependence
Brief Title: Treatment for Cannabis Withdrawal and Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Scripps Research Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Barbara J. Mason, Principal Investigator, The Scripps Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DA030988; 5R01DA030988-05 (NIH)
Record Dates: First submitted 2011-06-03; First posted 2012-06-05 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-03

CONDITIONS: Cannabis Dependence
MeSH Terms: conditions — Marijuana Abuse | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Drug (Active Comparator): 125mg/d aprepitant for 8 weeks given in conjunction with 8 weeks of manual-guided behavioral counseling.
  Interventions: Drug: Aprepitant; Behavioral: Manual-guided behavioral counseling
- Placebo pill (Placebo Comparator): Placebo pill daily for 8 weeks given in conjunction with 8 weeks of manual-guided behavioral counseling.
  Interventions: Drug: Placebo; Behavioral: Manual-guided behavioral counseling

INTERVENTIONS:
Drug: Aprepitant — 125mg/day for 8 weeks
  Other Names: Emend
  Arms: Active Drug
Drug: Placebo — 125mg/d placebo pill for 8 weeks
  Arms: Placebo pill
Behavioral: Manual-guided behavioral counseling — Standardized manual-guided behavioral counseling performed 1 time per week for 8 weeks in conjunction with study drug or placebo.
  Other Names: Manual-guided therapy

SUMMARY:
Cannabis is the most widely used illicit drug in the United States, and worldwide, with 1 in 10 users estimated to meet diagnostic criteria for cannabis dependence. Avoidance of withdrawal symptoms (e.g., disturbances in mood, sleep, and craving) is a common relapse precipitant. Cannabis use also impairs executive cognitive functions thereby increasing vulnerability to relapse and reducing the ability to benefit from behavioral therapy. There are no pharmacological treatments for cannabis dependence, despite the large number of afflicted individuals and the limitations of behavioral therapies which do not remediate withdrawal and are associated with high rates of treatment failure. The primary aim of this clinical trial is to evaluate the efficacy and safety of a novel neurokinin1 (NK1) receptor antagonist, aprepitant (Emend), (125mg/day), in outpatients with current cannabis dependence. The main hypothesis to be tested is to evaluate the relative efficacy of aprepitant 125 mg/d vs. placebo for reducing cannabis withdrawal symptoms in cannabis dependent outpatients, specifically anxiety, mood, craving and sleep.

DETAILED DESCRIPTION:
This study will be a Phase II, single-site, 8-week, randomized, double-blind, placebo-controlled, parallel group comparison of aprepitant (125 mg/d) or placebo. Subjects will be 100 outpatients seeking treatment for current cannabis dependence with no clinically significant medical or psychiatric disorders (including substance use disorders or a positive drug screen for substances other than cannabis or nicotine). All subjects will receive weekly manual-guided abstinence-oriented counseling to facilitate showing a drug effect above and beyond available therapies (Weeks 0-8). Research assessments of marijuana use and withdrawal and drug safety and tolerability will occur weekly through the treatment phase of the 8-week study. Post treatment follow-up assessments will occur at Weeks 9 and 12. Neuropsychological testing will occur at Weeks 0 and 4 and 8.

Specific Aim 1: To evaluate the relative efficacy of aprepitant 125 mg/d vs. placebo for reducing cannabis withdrawal symptoms in cannabis dependent outpatients, including anxiety, mood, craving and sleep symptoms.

Specific Aim 2: To evaluate the relative efficacy of aprepitant 125 mg/d vs. placebo for reducing marijuana use in cannabis dependent outpatients.

Specific Aim 3: To evaluate the relative efficacy of aprepitant 125 mg/d vs. placebo for reducing cannabis related impairments in executive functioning in cannabis dependent outpatients.

ELIGIBILITY:
Inclusion Criteria:

* Males or females from 18-70 years of age
* Meets DSM IV criteria for current cannabis dependence
* Seeking research-based outpatient treatment for cannabis dependence that involves daily oral medication
* Smoked MJ daily at least 25 days per month during the 90 days prior to randomization
* Current cannabis use verified by a positive urine test > 50 ng/ml
* At least a 2-year history of regular MJ use
* Willing and able to give informed consent

Exclusion Criteria:

* Abstinent from cannabis more than 2 days at the time of randomization
* Currently meets DSM IV criteria for dependence on substances, or has urine drug screen positive for substances, other than cannabis or nicotine
* Meets DSM IV criteria for a major AXIS I disorder other than cannabis and nicotine dependence,
* Active suicidal ideation
* Significant medical disorders that will increase potential risk or interfere with study participation,
* Females who are pregnant, nursing or who are sexually active with child-bearing potential and refuse to use a double-barrier method of birth control during the study and for up to 4 weeks after study termination
* Ongoing treatment with medications that may affect study outcomes,
* Use of CYP3A4 strong inhibitors (e.g., ketoconazole, itraconazole, nefazodone, troleandomycin, clarithromycin, ritonavir, nelfinavir) and CYP3A4 moderate inhibitors (e.g., diltiazem) within the 2 week period prior the study drug administration or within 5 half-lives of the respective medication, whichever is longer, until study conclusion.
* Consumption of grapefruit or grapefruit products from at least 2 weeks prior to study drug administration until study conclusion.
* Ongoing treatment with medications that are primarily metabolized by CYP3A4 and may have increased plasma concentrations when co-administered with aprepitant, such as pimozide, terfenadine, astemizole or cisapride or corticosteroids, as well as benzodiazepines including midazolam, alprazolam, and triazolam.
* Ongoing treatment with medications that are primarily metabolized by CYP2C9 (e.g., warfarin, tolbutamide).
* Use of drugs (e.g., rifampin, carbamazepine, phenytoin) or herbal supplements (e.g., St John's wort) that induce CYP3A4 activity and may result in reduced plasma concentrations of aprepitant and decreased efficacy of aprepitant.
* Inability to understand and/or comply with the provisions of the protocol and consent form.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Mason, Ph.D., Principal Investigator — The Scripps Research Institute
Locations (1):
- The Scripps Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study-related information — http://alcoholismmarijuanatreatment.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Aprepitant: 125mg/Day: 125mg/d aprepitant for 8 weeks given in conjunction with 8 weeks of manual-guided behavioral counseling.
- Matched Placebo: Matched Placebo daily for 8 weeks given in conjunction with 8 weeks of manual-guided behavioral counseling.
Period: Overall Study
Arm/Group | Aprepitant: 125mg/Day | Matched Placebo
Started | 32 | 38
Completed | 18 | 26
Not Completed | 14 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aprepitant: 125mg/Day | Matched Placebo | Total
Number analyzed (Participants) | 32 | 38 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.09 (10.62) | 30.50 (12.19) | 31.69 (11.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 23 | 29 | 52

OUTCOME MEASURES:

1. Primary Outcome: Change From Week 0 in Cannabis Use Using Urinary CN-THCCOOH Levels at Week 8
Description: Urinary THC/Cr ratio, also known as CN-THCCOOH (creatinine normalized tetrahydrocannabinol carboxylic acid), is a highly sensitive and specific quantitative analytic procedure to determine current marijuana metabolite levels in the urine as well as new marijuana use or abstinence. Gas chromatography mass spectrometric levels of 11-nor-9-carboxy-9-THC (THC-COOH), the primary marijuana metabolite, are normalized to the urine creatinine (CN) concentration to reduce the variability of drug measurement attributable to urine dilution. Negative values indicate decreased use. Change = (Week 8 value - Week 0 value).
Time Frame: Week 0 and Week 8
Population: Two participants in the matched placebo arm who completed the double blind portion of the trial were unable to be analyzed for change in Urinary CN-THCCOOH Level due to missing data at Week 0 and/or Week 8. One sample was missing source documentation while the other sample was too dilute to return a reliable measurement.
Measure: Mean (Standard Deviation); unit: ng/mg
Arm/Group | Aprepitant: 125mg/Day | Matched Placebo
Number analyzed (Participants) | 18 | 24
ng/mg | -334.21 (718.83) | -359.95 (1207.47)

ADVERSE EVENTS:
Arm/Group | Aprepitant: 125mg/Day | Matched Placebo
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/38
Other Adverse Events (participants affected / at risk) | 20/32 | 28/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aprepitant: 125mg/Day (N=32) | Matched Placebo (N=38)
Consipation (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 3
Fatigue (General disorders) | 0 | 3
Gastroenteritis viral (Infections and infestations) | 2 | 1
Nasopharyngitis (Infections and infestations) | 5 | 12
Joint injury (Injury, poisoning and procedural complications) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Dizziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 6 | 4
Somnolence (Nervous system disorders) | 3 | 3
Insomnia (Psychiatric disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No